CLINICAL TRIAL: NCT05914688
Title: A Bioequivalence Study of Subcutaneous Injections of LY3209590 in Two Formulations in Healthy Participants
Brief Title: A Study to Compare Two Formulations of LY3209590 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18310; I8H-MC-BDDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-14; First posted 2023-06-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Formulation; Bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY3209590 (Formulation 1) (Experimental): Single dose of LY3209590 as formulation 1 administered subcutaneously (SC).
  Interventions: Drug: LY3209590 (Formulation 1)
- LY3209590 (Formulation 2) (Experimental): Single dose of LY3209590 as formulation 2 administered SC.
  Interventions: Drug: LY3209590 (Formulation 2)

INTERVENTIONS:
Drug: LY3209590 (Formulation 1) — Administered SC.
  Arms: LY3209590 (Formulation 1)
Drug: LY3209590 (Formulation 2) — Administered SC.
  Arms: LY3209590 (Formulation 2)

SUMMARY:
The main purpose of this study is to compare the two formulations of LY3209590 in healthy participants. Study participants will be administered each formulation at separate study visits. Blood samples will be taken to compare how the body handles study drugs. The information about any adverse effects experienced will be collected and the tolerability of LY3209590 will also be evaluated.

Screening is required within 28 days prior to enrolment. For each participant, the total duration of the clinical trial will be about 184 days including screening.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are overtly healthy as determined by medical evaluation
* Have a body weight of 45 kilograms or more and body mass index (BMI) within the range of 18.5 to 35.0 kilograms per meter squared (kg/m²), inclusive
* Contraceptive use by participants should be consistent with local regulations

Exclusion Criteria:

* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, dermatological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have known allergies to LY3209590, related compounds, or any components of the formulation
* Have a history of multiple or severe allergic reactions or a history of severe anaphylactic reaction
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Are lactating or pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to the Last Time Point (AUC[0-tlast]) of LY3209590 | Predose up to 65 days post dose
  PK: AUC(0-tlast) of LY3209590
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3209590 | Predose up to 65 days post dose
  PK: AUC(0-∞) of LY3209590
PK: Maximum Observed Concentration (Cmax) of LY3209590 | Predose up to 65 days post dose
  PK: Cmax of LY3209590

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No